CLINICAL TRIAL: NCT04045691
Title: Encorafenib Plus Binimetinib in Patients With Locally Advanced, Unresectable or Metastatic BRAFV600-mutated Melanoma: a Multi-centric, Multinational, Prospective, Longitudinal, Non-interventional Study in Germany, Austria and Switzerland - BERING MELANOMA
Brief Title: Binimetinib Plus Encorafenib Real Life Investigation of Next Generation Melanoma Treatment
Acronym: BERING
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: Pierre Fabre Pharma Austria (Unknown); Pierre Fabre Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PFO-2019-1921
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Melanoma Stage IV; Melanoma Stage III
Keywords: BERING; Encorafenib; Binimetinib
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Encorafenib — Observation of real-life treatment with encorafenib and binimetinib
Drug: Binimetinib — Observation of real-life treatment with encorafenib and binimetinib

SUMMARY:
BERING-MELANOMA - designed as a prospective, longitudinal, non-interventional study - investigates real-world effectiveness, quality of life, safety and tolerability of encorafenib plus binimetinib in unresectable advanced or metastatic BRAF(Rapidly Accelerated Fibrosarcoma isoform B)-V600-mutant malignant melanoma after commercial availability of these two products in Germany, Austria and Switzerland. The study focusses on the documentation of the first and second line setting (i.e. after one line of prior checkpoint inhibition) by documenting patients treated according to the SmPC (Summary of Product Characteristics).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient with regard to the pseudonymized documentation as well as the transfer and processing of his/her data within the study and the ADOREG [Cancer Registry of German Working Group of Dermato-Oncology] registry (data transfer to ADOREG registry only for patients from German sites);
* Legally capable male or female patient ≥ 18 years of age (no upper limit);
* Decision was taken to treat the patient with encorafenib plus binimetinib in accordance with the current SmPC [Summary of Product Characteristics] and by prescription; this decision was taken prior to and independent from the inclusion into the study;
* Treatment with encorafenib plus binimetinib has been started ≤ 6 months prior to providing written informed consent for this study or is planned to be started in the near future;
* Unresectable advanced or metastatic malignant melanoma with BRAF [Rapidly Accelerated Fibrosarcoma isoform B] V600 mutation;
* Treatment-naive or after one prior line of checkpoint inhibitor treatment (anti-CTLA4 [Cytotoxic T-Lymphocyte Antigen-4] and/or anti-PD(L)1 [Programmed cell Death protein 1]) in the unresectable advanced or metastatic setting.

Exclusion Criteria:

* Previous treatment with a BRAF- and/or MEK [Mitogen-Activated Protein/Extracellular-signal Regulated Kinase]- inhibitor except for:

  -- prior adjuvant treatment with BRAF+MEK-inhibitor combination therapy that ended > 6 months prior start of Encorafenib/Binimetinib treatment;
* More than one prior line of checkpoint inhibitor treatment in the unresectable advanced or metastatic setting;
* Any previous chemotherapeutic treatment of the melanoma disease;
* Presence of any contraindication with regard to the encorafenib-binimetinib-treatment as specified in the corresponding SmPCs;
* Current or upcoming participation in an interventional clinical trial;
* Current or upcoming systemic treatment of any other tumor than melanoma;
* Prisoners or persons who are compulsorily detained (involuntarily incarcerated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with unresectable advanced or metastatic BRAFV600-mutant malignant melanoma, with a decision to receive targeted treatment with Encorafenib/Binimetinib according to the current SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | At 12 months after start of treatment
  Progression-free survival rate

SECONDARY OUTCOMES:
Patient and disease profiles at start of treatment with encorafenib plus binimetinib | Baseline
  Demographic and disease characteristics
Type of treatments before and after encorafenib plus binimetinib | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Treatment sequence prior to and after encorafenib plus binimetinib; by documenting pre-treatments with adjuvant therapy and systemic therapy in palliative setting; and by documenting subsequent systemic treatment lines after administration of encorafenib plus binimetinib
Sequence of treatments before and after encorafenib plus binimetinib | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Treatment sequence prior to and after encorafenib plus binimetinib; by documenting pre-treatments with adjuvant therapy and systemic therapy in palliative setting; and by documenting subsequent systemic treatment lines after administration of encorafenib plus binimetinib
Characteristics of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Evaluation of reason for treatment selection (efficacy, safety profile, quality of life, patients preference, physician's preference, comorbidities, other)
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Further progression-free survival parameters
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Time-to-progression
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Best observed tumor response
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Overall response rate
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Duration of response
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Disease control rate
Effectiveness of treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Duration of disease control
Effectiveness of treatment with encorafenib plus binimetinib | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Overall survival
Patient reported outcomes during treatment with encorafenib plus binimetinib - evaluated with EORTC QLQ C-30 | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  EORTC QLQ C-30 questionnaires (European Organisation for Research and Treatment of Cancer Quality of Life C-30 questionnaires) to assess quality of life of cancer patients; comprises 30 items, 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms.
Patient reported outcomes during treatment with encorafenib plus binimetinib evaluated with WPAI | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  WPAI questionnaires (Work Productivity and Activity Impairment questionnaires). The following questions ask about the effect of patients melanoma on the ability to work and perform regular activities.
  1. Are you currently employed (working for pay)?
  2. During the past seven days, how many hours did you miss from work because of problems associated with your melanoma?
  3. During the past seven days, how many hours did you miss from work because of any other reason?
  4. During the past seven days, how many hours did you actually work?
  5. During the past seven days, how much did your melanoma affect your productivity while you were working?
  6. During the past seven days, how much did your melanoma affect your ability to do your regular daily activities, other than work at a job?
Patient reported outcomes during treatment with encorafenib plus binimetinib evaluated with CTSQ | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  CTSQ questionnaires (Cancer Therapy Satisfaction Questionnaire) to assess patients' opinions and feelings concerning their cancer therapy and associated adverse events:
  1. Questions to patients thoughts about cancer therapy (IV/pills). Scale: [Always, Most of the time, Some-times, Rarely, Never];
  2. Questions to patients satisfaction with the most recent cancer therapy (IV/pills):
     1. Scale reg. benefit: [Much better than my expectations Somewhat better than my expectations, Met my expectations, Somewhat worse than my expectations, Much worse than my expectations];
     2. Scale reg. side effects: [Much better than I expected, Somewhat better than I expected, Exactly as I expected, Somewhat worse than I expected, Much worse than I expected];
     3. Scale reg. satisfaction: [Very satisfied, Satisfied, Neither satisfied nor dissatisfied, Dissatisfied, Very dissatisfied];
     4. Scale reg. choice of therapy: [Yes, definitely, Probably Yes, I don't know, Probably not, Definitely not]
Physicians' satisfaction with regard the treatment with encorafenib plus binimetinib | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  Physicians' satisfaction questionnaires (measuring Physician's Satisfaction with regard to Effictiveness and Safety, as well as Physician's Overall Treatment Satisfaction) using the following scale construct:
  1. Physician's Satisfaction with regard to Efficiency
  2. Physician's Satisfaction with regard to Safety
  3. Physician's Overall Treatment Satisfaction
  Scale:
  * very dissatisfied
  * dissatisfied
  * moderately satisfied
  * satisfied
  * very satisfied
Safety and tolerability of treatment with encorafenib plus binimetinib - Adverse events and adverse reactions including time to onset and time to resolution | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Number of patients with Adverse Events and maximum grade per patient, Adverse Drug Reactions, Adverse Drug Reactions grade 3/4, Serious Adverse Events, Serious Adverse Drug Reactions.
Prognostic factors | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Influence of prognostic factors on quality of life outcome parameters
Prognostic factors | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Influence of prognostic factors on effectiveness
Prognostic factors | Complete observation time-frame (the total observation period of this study will amount to 90 months).
  Influence of prognostic factors on safety
Treatment duration | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  From date of first treatment (encorafenib or binimetinib, whichever occurs first) until date of last treatment (encorafenib or binimetinib, whichever occurs last)
Treatment dose intensity | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  From date of first treatment (encorafenib or binimetinib, whichever occurs first) until date of last treatment (encorafenib or binimetinib, whichever occurs last)
Number of treatment interruptions | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  From date of first treatment (encorafenib or binimetinib, whichever occurs first) until date of last treatment (encorafenib or binimetinib, whichever occurs last)
Duration of treatment interruptions | From start to end of treatment (anticipated median treatment duration ca. 12 months)
  From date of first treatment (encorafenib or binimetinib, whichever occurs first) until date of last treatment (encorafenib or binimetinib, whichever occurs last)

CONTACTS AND LOCATIONS:
Locations (59):
- Austria (9):
  - 11, Graz
  - 13, Innsbruck
  - 14, Klagenfurt
  - 10, Linz
  - 3, Linz
  - 12, Salzburg
  - 22, Vienna
  - 53, Vienna
  - 23, Wiener Neustadt
- Germany (42):
  - 45, Ahaus
  - 8, Aschaffenburg
  - 56, Augsburg
  - 51, Berlin
  - 27, Bremerhaven
  - 1, Buxtehude
  - 43, Chemnitz
  - 34, Donauwörth
  - 49, Dresden
  - 47, Duisburg
  - 40, Erfurt
  - 20, Essen
  - 9, Gera
  - 28, Giessen
  - 42, Goslar
  - 59, Göttingen
  - 19, Hamburg
  - 21, Hanover
  - 2, Heidelberg
  - 33, Karlsruhe
  - 39, Kiel
  - 29, Landshut
  - 44, Leipzig
  - 30, Ludwigshafen
  - 4, Lübeck
  - 46, Magdeburg
  - 15, Mainz
  - 5, Mannheim
  - 57, Marburg
  - 6, Minden
  - 31, München
  - 7, München
  - 16, Münster
  - 35, Münster
  - 18, Nuremberg
  - 50, Regensburg
  - 41, Schorndorf
  - 17, Schwerin
  - 48, Stolberg
  - 55, Trier
  - 54, Tübingen
  - 32, Zwickau
- Switzerland (8):
  - 52, Bellinzona, Canton Ticino
  - 38, Aarau
  - 37, Bern
  - 24, Chur
  - 36, Lausanne
  - 58, Lucerne
  - 26, Winterthur
  - 25, Zurich

IPD SHARING:
Plan to Share IPD: No